CLINICAL TRIAL: NCT03397628
Title: FIFA 11 for Health in Europe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Peter Krustrup, Professor, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Purpose: Prevention
Other Study IDs: FIFA11fh
Record Dates: First submitted 2016-09-23; First posted 2018-01-12 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Health Knowledge, Attitudes, Practice
MeSH Terms: conditions — Behavior | interventions — Health

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention)
- Intervention (Experimental)
  Interventions: Other: FIFA 11 for health

INTERVENTIONS:
Other: FIFA 11 for health
  Arms: Intervention

SUMMARY:
Proposed action: To investigate the effect of an innovative and easily implementable football-based health education programme on well-being, self-esteem, health knowledge and physical fitness for 10-12-year old school children. The programme has been running in 22 countries in Africa and South America and is now being adapted to the Western World. The first step was to run a pilot implementation for more than 600 school children in Copenhagen, Frederiksberg, Roskilde and Frederikssund in the school year 2015-2016. From august 2016 to a nationwide implementation for 30,000 school children is started in Denmark and The Faroe Islands.

DETAILED DESCRIPTION:
Proposed action: To investigate the effect of an innovative and easily implementable football-based health education programme on well-being, self-esteem, health knowledge and physical fitness for 10-12-year old school children. The programme has been running in 22 countries in Africa and South America and is now being adapted to the Western World. The first step was to run a pilot implementation for more than 600 school children in Copenhagen, Frederiksberg, Roskilde and Frederikssund in the school year 2015-2016. From august 2016 to a nationwide implementation for 30,000 school children is started in Denmark and The Faroe Islands. The programme is developed and implemented in a close collaboration between the University of Southern Denmark, University of Copenhagen, The Danish Football Association and the international football association FIFA, and the ambitious scope of the project is to continue this collaboration in a large-scale implementation involving up to 1 million children in up to 30 Western Countries.

As in Africa and South America FIFA is providing all equipment for the programme, including footballs, cones, bibs, training manuals etc. FIFA and the Danish FA have employed a co-funded national project leader in Denmark for a 3-year period, starting August 2015.

The University of Southern Denmark and the Danish FA is responsible for the training manuals, coaching courses for school teachers and the research related the nationwide implementation.

Main project activities: The FIFA 11 for Health in Denmark programme is being delivered 30,000 school children aged 10-12 (5th grade pupils) in the nationwide implementation phase. The programme is being delivered by two school teachers (one female and one male teacher) in each of the schools, and includes two weekly 45-min sessions per week over an 11-week period. The football-based health education programme incorporates fun, joyful and social small-sided games and pair-exercises along with specific focus on one important health message in week. Girls and boys will play together, and the exercises are conducted so that all the children will have a high involvement, success rate and intensity, also the unfit, obese, and non-sport club active. At the same time the exercises are constructed with special focus on how to be a good friend and a team player, how to demonstrate empathy and skill in helping others both individually and as a group, and how to avoid bullying and how to think positively. The 11 health messages cover the most important and prominent health challenges of the Western World, including importance social wellbeing, mental health, physical activity, diet, hygiene and risk-behavior such as abuse of alcohol and drugs.

ELIGIBILITY:
Inclusion Criteria:

* Healthy

Exclusion Criteria:

* Disabilities

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20000 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Health Knowledge | up to 2 yrs
  questionnaire

SECONDARY OUTCOMES:
Fitness | up to 2 yrs
  physical testing
Well-being | up to 2 yrs
  questionnaire
Cognitive function | up to 2 yrs
  Cogstate test battery

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern Denmark, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No